CLINICAL TRIAL: NCT06510270
Title: Targeting Epicardial Adipose Tissue in Heart Failure with Preserved Ejection Fraction: Exploring the Dapagliflozin Connection
Brief Title: Dapagliflozin in Reducing Epicardial Adipose Tissue in Heart Failure with Preserved Ejection Fraction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Aml Soliman, Lecturer of cardiology, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 865/11/23
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure with Preserved Ejection Fraction
Keywords: HFpEF, Dapagliflozin, epicardial adipose tissue
MeSH Terms: interventions — dapagliflozin; Sodium Potassium Chloride Symporter Inhibitors; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Symptomatic heart failure (Active Comparator): Patients with clinical manifictations of heart failure but preserved ejection fraction by echocardiography.
  Interventions: Drug: Dapagliflozin 10 mg once daily; Drug: Loop diuretics; Drug: Treatments of associated co-morbidities (e.g Anti-hypertensive, oral hypoglycemic)
- Asymptomatic Diastolic dysfunction (Placebo Comparator): Patients with diastolic dysfunction grade II or more by Echocardiography but with out any heart failure manifictation.
  Interventions: Drug: Treatments of associated co-morbidities (e.g Anti-hypertensive, oral hypoglycemic)

INTERVENTIONS:
Drug: Dapagliflozin 10 mg once daily — Dapagliflozin 10 mg once daily will be given to all patients in symptomstic heart failure group
  Arms: Symptomatic heart failure
Drug: Loop diuretics — Loop diuretics (IV or orally) will be given to all patients in symptomatic heart failure group
  Arms: Symptomatic heart failure
Drug: Treatments of associated co-morbidities (e.g Anti-hypertensive, oral hypoglycemic) — Treatment of associated co-morbidities will be given to both arms (group) such as anti-hypertensive (B blockers, ACIE, ARBS, CA channel blockers, Diuretics), oral hypoglycemic (Metformins, sulfonyl urea,.......)

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is becoming the most common cause of heart failure worldwide, in part, driven by a rising prevalence of obesity.

Although generalized and visceral adiposity is important in the pathogenesis of obesity-related HFpEF, there is increasing recognition of the potential role of epicardial adipose tissue (EAT) in disease pathogenesis. EAT is metabolically active tissue located directly on the surface of the myocardium underneath the visceral pericardium. By virtue of its anatomical interface with the heart and the lack of fascial separation between the underlying myocardium and epicardial fat, locally secreted adipokines directly bathe the surface of the heart and result in underlying myocardial remodeling.

Its position on the surface of the myocardium allows EAT to directly contribute to an increase in total heart size with stretch of the pericardium and results in relative pericardial restraint with constrictive physiology.

EAT is most commonly measured by echocardiography in the parasternal long axis view perpendicular to the right ventricle (RV) to quantify epicardial fat thickness and this has been correlated with worse haemodynamic derangements and adverse outcomes in HFpEF.

Alternatively, cardiac MRI or CT can provide a more complete volumetric assessment of epicardial fat volume and has also demonstrated associations with adverse outcomes and functional metrics in most but not all HFpEF studies.

Very little is understood about the impact of medical modulation of epicardial fat in HFpEF. The first proven agents to improve heart failure hospitalization and quality of life in HFpEF are the sodium-glucose cotransporter-2 inhibitors (SGLT2i) Although the mechanisms of benefit of these drugs are uncertain, they have demonstrated a reduction in epicardial fat despite only minimal weight loss suggesting a direct lipolytic effect on epicardial fat. The use of SGLT2i has also been associated with reduced incident AF, which may, in part, be due to the reduction in epicardial fat. The diuretic effect of SGLT2i may facilitate a reduction in plasma volume and mechanistic studies have shown that they also promote ventricular mass regression, which may cumulatively decrease pericardial restraint.

By this work we aims To determine whether the addition of 10 mg of Dapagliflozin to a patient with HFPEF can lead to a decrease in epicardial adipose tissue volume, which is a new approach to managing HFPEF or not.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Patients with established diagnosis of HFpEF: (1. Signs and Symptoms of Heart Failure. 2. Preserved Ejection Fraction (EF): EF greater than or equal to 50% is generally considered preserved. 3.Echo-cardiography: Evidence of left ventricular hypertrophy (LVH) or Evidence of diastolic dysfunction, such as impaired relaxation or increased stiffness of the left ventricle. 4.Elevated Natriuretic Peptides: serum N-terminal pro-B type natriuretic peptide (NT-proBNP) ≥400 pg/mL or brain natriuretic peptide ≥100 pg/mL can support the diagnosis of HFpEF in the presence of symptoms and other findings).
3. BMI >27Kg/m2.
4. Adequate follow-up: Participants must be willing and able to comply with the study protocol and follow-up requirements.

Exclusion Criteria:

* 1. Age <18 years. 2. Type 1 diabetes: Exclude individuals with type 1 diabetes, as dapagliflozin is primarily used for type 2 diabetes management.

  3. Significant renal impairment: Exclude participants with severe renal impairment or end-stage renal disease.

  4. Severe hepatic impairment: Exclude participants with severe hepatic dysfunction.

  5. Pregnancy or breastfeeding: Exclude pregnant or lactating individuals. 6. Patients who underwent Bariateric surgery. 7. BMI<27Kg/m2. 8. Other serious medical conditions: Exclude participants with serious medical conditions that could interfere with the study or confound the results (e.g., cancer, severe infections).

  9. Inability to comply: Exclude participants who are unable or unwilling to comply with the study procedures and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Epicardial adipose tissue volume | from enrollment (before stsrting dapagliflozin) to 6 month (while still on dapagliflozin)
  epicardial adipose tissue volume (gm) will be measured by using CMR before starting Dapagliflozin in sympotomatic heart failure group and 6 months latter. In asymptomatic diastolic dysfunction CMR will be performed at enrollment and 6 month latter

SECONDARY OUTCOMES:
Change in Body mass index | At enrollement till 6 months latter
  body mass index (kg/m2) will be measured at enrollment for both groups and 6 month latter at the end of the study
Recurrent hospital admission by heart failure | From enrollement till 6 months latter
  Number of recurrent hospital admission by heart failure for each participant from enrollment till th end of study (6 month latter) will be recorded
Cardio-vascular mortality | From enrollement till 6 months latter
  Cardiovascular mortality rate (due to stroke or MI) will be measured for both groups

IPD SHARING:
Plan to Share IPD: Undecided